CLINICAL TRIAL: NCT02588625
Title: A Double-Blinded Study to Evaluate the Safety, Tolerability, and Efficacy of BMS-986020 Versus Placebo in Diffuse Cutaneous Systemic Sclerosis (dcSSc)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM136-132
Record Dates: First submitted 2015-10-26; First posted 2015-10-28 (Estimated); Last update posted 2016-07-22 (Estimated); Status verified 2016-07

CONDITIONS: Scleroderma
MeSH Terms: conditions — Scleroderma, Diffuse

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Part A - BMS-986020 (Experimental): BMS-986020 or Placebo tablets specified dose on specified days
  Interventions: Drug: BMS-986020; Other: Placebo
- Part B - BMS-986020 (Experimental): BMS-986020 or Placebo tablets specified dose on specified days
  Interventions: Drug: BMS-986020; Other: Placebo

INTERVENTIONS:
Drug: BMS-986020
Other: Placebo

SUMMARY:
This is a two part study.

The purpose of Part A is to determine if BMS-986020 is effective in treatment of diffuse cutaneous systemic sclerosis using one dose of BMS-986020.

The purpose of Part B is to determine if BMS-986020 is effective in treatment of diffuse cutaneous systemic sclerosis using two different doses of BMS-986020.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Diagnosis of diffuse cutaneous systemic sclerosis for 60 months or less
* Men and women ≥ 18 years of age
* Ability to comply with birth control requirements
* Certain immunosuppressive agents are permitted

Exclusion Criteria:

* Limited cutaneous systemic sclerosis or sine scleroderma
* Active ulcers on fingers
* Pulmonary arterial hypertension
* Any gastrointestinal surgery that may impact absorption of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-02; Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Part A - Change in modified Rodnan skin score (mRSS) | Week 24
Part B - Change in modified Rodnan skin score (mRSS) | Week 48

SECONDARY OUTCOMES:
Part A: Change in physical function based on health assessment questionnaire-disability index from baseline at specified timepoints (HAQ-DI) | Week 4, 12 and 24
Part A: Change in percent predicted forced vital capacity (FVC) from baseline at specified time points | Week 4, 12 and 24
Part A: Proportion of subjects with ≥ 20%, 40%, or 60% change in mRSS from baseline at specified time points | Week 4, 12 and 24
Part A: Change in subject's global assessment on a visual analog scale (VAS) from baseline at specified time points | Week 4, 12 and 24
Part A: Change in physician's global assessment on a visual analog scale (VAS) from baseline at specified time points | Week 4, 12 and 24
Part A: Safety as measured by the frequency of deaths, SAEs, drug related AEs, AEs leading to discontinuation as well as marked abnormalities in clinical laboratory tests, vital sign measurements, ECGs, physical examinations | up to Month 3 of the Follow-Up
  Serious adverse event (SAE), Adverse event (AE)
Part A: Tolerability as measured by the frequency of deaths, SAEs, drug related AEs, AEs leading to discontinuation as well as marked abnormalities in clinical laboratory tests, vital sign measurements, ECGs, physical examinations | up to Month 3 of the Follow-Up
Part B: Change in physical function based on health assessment questionnaire-disability index (HAQ-DI) | Week 48
Part B: Change in percent predicted forced vital capacity | Week 48
Part B:Proportion of subjects with ≥ 20%, 40%, or 60% change in mRSS from baseline at specified time points | Week 4, 12, 24, 36, and 48
Part B: Proportion of subjects with > 10% absolute decline in % FVC | Week 48
Part B:Proportion of subjects with % FVC change > 0 | Week 48
Part B: Change in quantitative lung fibrosis (QLF) score on High resolution CT (HRCT) from baseline at specified time points | Week 48
Part B: Change in subject's global assessment on a visual analog scale (VAS) from baseline at specified time points | Week 4, 12, 24, 36, and 48
Part B: Change in physician's global assessment on a visual analog scale (VAS) from baseline at specified time points | Week 4, 12, 24, 36, and 48
Part B: Change in health-related quality of life (HRQOL) using Patient Reported Outcomes Measurement Information System (PROMIS)-29 score from baseline at specified time points | Week 4, 12, 24, 36, and 48
Part B: Safety as measured by the frequency of deaths, SAEs, drug related AEs, AEs leading to discontinuation as well as marked abnormalities in clinical laboratory tests, vital sign measurements, ECGs, physical examinations | up to Month 3 of the Follow-Up
Part B: Tolerability as measured by the frequency of deaths, SAEs, drug related AEs, AEs leading to discontinuation as well as marked abnormalities in clinical laboratory tests, vital sign measurements, ECGs, physical examinations | up to Month 3 of the Follow-Up

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (24):
- United States (16):
  - Local Institution, Scottsdale, Arizona
  - Local Institution, Los Angeles, California
  - Local Institution, Stanford, California
  - Local Institution, Aurora, Colorado
  - Local Institution, Washington D.C., District of Columbia
  - Local Institution, Chicago, Illinois
  - Local Institution, Baltimore, Maryland
  - Local Institution, Boston, Massachusetts
  - Local Institution, Ann Arbor, Michigan
  - Local Institution, New Brunswick, New Jersey
  - Local Institution, Albany, New York
  - Local Institution, New York, New York
  - Local Institution, Cleveland, Ohio
  - Local Institution, Pittsburgh, Pennsylvania
  - Local Institution, Charleston, South Carolina
  - Local Institution, Houston, Texas
- Canada (2):
  - Local Institution, Hamilton, Ontario
  - Local Institution, London, Ontario
- Poland (5):
  - Local Institution, Bydgoszcz
  - Local Institution, Lublin
  - Local Institution, Poznan
  - Local Institution, Szczecin
  - Local Institution, Warsaw
- Local Institution, London, Greater London, United Kingdom

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx